CLINICAL TRIAL: NCT00920140
Title: An Open-Label, Dose-Escalation, Phase I/II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of the MEK Inhibitor GSK1120212 in Subjects With Relapsed or Refractory Leukemias
Brief Title: Open-label Study to Evaluate the Safety, PK, and PD of MEK Inhibitor GSK1120212 in Subjects With Relapsed or Refractory Leukemias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111759
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Cancer
Keywords: Oncology, GSK1120212, MEK inhibitor, hematological malignancies, AML; CMML; MDS
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Leukemia, Myeloid, Acute | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (Experimental): The proposed treatment schedule of GSK1120212 is continuous daily dosing. At the initiation of dosing, a loading dose will be given prior to starting continuous dosing (maintenance dose).
  Alterations to the dose and schedule will be based on emerging PK, PD, and tolerability data. The goal will be to define a regimen that is well tolerated and provides adequate PK and PD. This will be the recommended Phase II schedule.
  Interventions: Drug: GSK1120212
- Phase II (Experimental): A dose determined by Phase I to further evaulate the safety profile, PK, PD, and clinical activity of GSK1120212.
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Starting dose based on GSK protocol MEK111054 and then dose escalation based on Dose Limiting Toxicities per protocol.
  Arms: Phase I
Drug: GSK1120212 — Dose will be maximum tolerated dose based on Phase I results.
  Arms: Phase II

SUMMARY:
MEK111759 is a dose-escalation, Phase I/II, open-label study to determine the recommended dose and regimen for the orally administered MEK inhibitor GSK1120212 in subjects with relapsed or refractory leukemias. The recommended dose and regimen will be selected based on the safety, pharmacokinetic, and pharmacodynamic profiles. This study will identify the maximum tolerated and recommended Phase II doses using a dose-escalation procedure. Dose escalations will continue based on predefined parameters until a maximum tolerated dose is established. In Phase II, the clinical efficacy of GSK1120212 in subjects with relapsed or refractory leukaemias (AML, MDS or CMML) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Phase I
* Written informed consent provided.
* 18 years old or older.
* Subjects must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable remission. Subjects with poor-risk myelodysplasia (MDS) and chronic melomonocytic leukemia (CMML) are also eligible. Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML), acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Subjects with agnogenic myeloid metaplasia (AMM) are also eligible. Subjects with a haematological malignancy associated with human immunodeficiency virus (HIV) infection or solid organ transplant are NOT eligible.
* Subjects who have previously received an autologous stem cell transplant are allowed if a minimum of three months has elapsed from the time of transplant (T0) and the subject has recovered from transplant-associated toxicities prior to the first dose of GSK1120212.
* Subjects with a history of allogeneic stem cell transplant are eligible for study participation provided the following eligibility criteria are met: transplant was greater than 100 days prior to study enrolment, subject has not taken immunosuppressive medications (per protocol) for at least 1 month, no signs or symptoms of graft versus host disease other than Grade 1 skin involvement, no active infection, subject meets the remainder of the eligibility criteria outlined in this protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
* Life expectancy of at least four weeks.
* Able to swallow and retain oral medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol.
* Female subjects must be of non-childbearing potential as listed in the protocol or using a contraception method listed in the protocol.
* Calcium Phosphate Product less than or equal to 4.0 mmol (squared)/L (squared) or 50mg (squared)/dL (squared).
* Subjects must have adequate organ function as specified in the protocol.
* Phase II
* Confirmed diagnosis of one of the following: Relapsed or refractory acute myeloid leukemia (AML), Secondary AML including AML arising from antecedent hematologic diseases (e.g., myelodysplastic syndrome, myeloproliferative disorders, or therapyrelated AML), CMML, or MDS.

Cohorts 1: RAS Positive AML/MDS Cohort 2: Wild Type AML/MDS/CMML Cohort 3: RAS Positive CMML

Exclusion Criteria:

* Phase I
* Currently receiving cancer therapy as specified in the protocol.
* Received corticosteroids or imatinib within 24h of GSK1120212 administration.
* Received gemtuzumab ozogamicin (myelotarg) within two weeks of GSK1120212 adminstration.
* Received an investigational anti-cancer drug within four weeks or five half-lives, whichever is shorter of GSK1120212 administration, as specified in the protocol.
* Received major surgery, radiotherapy, or immunotherapy within four weeks of GSK1120212 administration.
* Received chemotherapy regimens with delayed toxicity within the last four weeks (six weeks for prior nitrosourea or mitomycin C). Received chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last two weeks.
* Received a MEK inhibitor.
* Current use of a prohibited medication per protocol.
* Current use of warfarin. Low molecular weight heparin and prophylactic low-dose warfarin are permitted per protocol.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* History of RVO.
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein thrombosis.
* Intraocular pressure greater than 21mm Hg as measured by tonography.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Condition that in the investigator's opinion would jeopardize compliance with the protocol.
* Symptomatic or untreated central nervous system involvement by the hematologic malignancy, including primary CNS lymphoma. Subjects who were previously treated for CNS involvement, and are asymptomatic without anti-epileptic medications for at least two months are eligible.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Unresolved toxicity greater than Grade 1 from previous anti-cancer therapy except alopecia (if applicable) unless agreed to by a GSK Medical Monitor and the investigator.
* QTc interval greater than 480 msecs.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, dimethyl sulfoxide (DMSO), or excipients (See Section 3.10). (To date there are no known FDA approved drugs chemically related to GSK1120212).
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (15):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Bornx, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- France (5):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Toulouse
- Germany (6):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Phase I/II study. Phase I is a dose escalation phase in participants with relapsed or refractory leukaemias to identify the recommended dose of GSK1120212 for Phase II. Phase II further evaluates the safety and efficacy of the recommended dose.
Groups:
- GSK1120212 < 2 mg OD: Participants with relapsed or refractory leukemias received either GSK1120212 3 milligrams (mg) loading dose (LD) followed by 1 mg once daily (OD) (3/1 mg LD/OD), or 1 mg OD as a continuous dose.
- GSK1120212 2 mg OD: Participants with relapsed or refractory leukemias received GSK1120212 2 mg OD as a continuous dose.
- Cohort 1: AML/MDS With RAS Mutation: Participants with relapsed or refractory acute myeloid leukemia (AML) or myelodysplasia (MDS) with rat sarcoma (RAS) mutation received GSK1120212 2 mg OD as a continuous dose.
- Cohort 2: AML/MDS/CMML With RAS wt/Unknown: Participants with relapsed or refractory AML or MDS or chronic myelomonocytic leukemia (CMML) with RAS wild type (wt) or unknown mutation received GSK1120212 2 mg OD as a continuous dose.
- Cohort 3: CMML With RAS Mutation: Participants with relapsed or refractory CMML with RAS mutation received GSK1120212 2 mg OD as a continuous dose.
Period: Phase 1 (Dose Escalation)
Arm/Group | GSK1120212 < 2 mg OD | GSK1120212 2 mg OD | Cohort 1: AML/MDS With RAS Mutation | Cohort 2: AML/MDS/CMML With RAS wt/Unknown | Cohort 3: CMML With RAS Mutation
Started | 5 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Period: Phase 2
Arm/Group | GSK1120212 < 2 mg OD | GSK1120212 2 mg OD | Cohort 1: AML/MDS With RAS Mutation | Cohort 2: AML/MDS/CMML With RAS wt/Unknown | Cohort 3: CMML With RAS Mutation
Started | 0 | 0 | 50 | 22 | 11
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 50 | 22 | 11
Not completed — Adverse Event | 0 | 0 | 14 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 29 | 14 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 3 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1120212 <2 mg OD: Participants with relapsed or refractory leukemias received either GSK1120212 3 milligrams (mg) loading dose (LD) followed by 1 mg once daily (OD) (3/1 mg LD/OD), or 1 mg OD as a continuous dose.
- Cohort 1: AML/MDS With RAS Mutation: Participants with relapsed or refractory AML or MDS with RAS mutation received GSK1120212 2 mg OD as a continuous dose.
- Cohort 2: AML/MDS/CMML With RAS wt/Unknown: Participants with relapsed or refractory AML or MDS or CMML with RAS wt or unknown mutation received GSK1120212 2 mg OD as a continuous dose.
- Total: Total of all reporting groups
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD | Cohort 1: AML/MDS With RAS Mutation | Cohort 2: AML/MDS/CMML With RAS wt/Unknown | Cohort 3: CMML With RAS Mutation | Total
Number analyzed (Participants) | 5 | 9 | 50 | 22 | 11 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (15.71) | 60.2 (15.86) | 65.6 (10.71) | 59.6 (18.89) | 67.7 (6.87) | 64.2 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 22 | 7 | 6 | 41
  Male | 1 | 7 | 28 | 15 | 5 | 56
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 5 | 2 | 0 | 8
  White - White/Caucasian/European Heritage | 4 | 9 | 40 | 18 | 9 | 80
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 1 | 2
  Asian - Japanese Heritage | 0 | 0 | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0 | 1 | 0 | 1
  Missing | 0 | 0 | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) by Dose
Description: An AE is any untoward medical occurrence in a participant (par.) or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: All Treated Population: all participants who received at least one dose of study medication. Safety data was evaluated based on this population. One Phase 2 par. was incorrectly dosed (received <2 mg [0.5 mg]); thus, 6 par. receiving GSK1120212 <2 mg OD were analyzed.
Measure: Number; unit: Participants
Groups:
- GSK1120212 <2 mg OD: Participants with relapsed or refractory leukemias received either GSK1120212 3 mg LD followed by 1 mg OD (3/1 mg LD/OD), or 1 mg OD as a continuous dose.
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  Any AE | 6 | 91
  Any SAE | 2 | 64

2. Primary Outcome: Number of Participants With a Change From Baseline Grade to Grade 3 and 4 for the Indicated Hematology Parameters by Dose
Description: Hematology and clinical chemistry data were summarized according to National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade, version 3.0. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. Hematology tests where the toxicity grade is defined by NCI-CTCAE includes hemoglobin, international normalized ratio (INR), lymphocytes, total neutrophils, platelet count, and partial thromboplastin time (PTT). Participants with missing baseline grades were assumed to have a baseline grade of 0. Only those participants (par.) with laboratory values for worst-case on-therapy (defined as the worst shift that occurred at any time during the treatment period) are presented.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: All Treated Population (ATP). Only those par. available at the specified time points were analyzed. Different par. may have been analyzed for different parameters; the overall number analyzed reflects everyone in the ATP. One Phase 2 par. was incorrectly dosed (received <2 mg [0.5 mg]); thus, 6 par. receiving GSK1120212 <2 mg OD were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  Hemoglobin (Low), Grade 3, n=6, 91 | 3 | 28
  Hemoglobin (Low), Grade 4, n=6, 91 | 0 | 7
  INR (High), Grade 3, n=6, 75 | 0 | 0
  INR (High), Grade 4, n=6, 75 | 0 | 0
  Lymphocytes (Low), Grade 3, n=6, 90 | 0 | 12
  Lymphocytes (Low), Grade 4, n=6, 90 | 0 | 7
  Total Neutrophils (Low), Grade 3, n=6, 89 | 1 | 4
  Total Neutrophils (Low), Grade 4, n=6, 89 | 1 | 21
  Platelet count (Low), Grade 3, n=6, 91 | 0 | 5
  Platelet count (Low), Grade 4, n=6, 91 | 1 | 28
  PTT (High), Grade 3, n=5, 75 | 0 | 1
  PTT (High), Grade 4, n=5, 75 | 0 | 0
  White Blood Cell count (Low), Grade 3, n=6, 91 | 1 | 13
  White Blood Cell count (Low), Grade 4, n=6, 91 | 0 | 15

3. Primary Outcome: Number of Participants With a Change From Baseline Grade to Grade 3 and 4 for the Indicated Clinical Chemistry Parameters by Dose
Description: Hematology and clinical chemistry data were summarized according to NCI-CTCAE grade, version 3.0. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. Clinical chemistry tests where the toxicity grade is defined by NCI-CTCAE includes albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase (AST), total bilirubin, calcium, creatinine, glucose, bicarbonate, potassium, magnesium, sodium, and phosphorus. Participants with missing Baseline grades were assumed to have a Baseline grade of 0. Only those participants (par.) with laboratory values for worst-case on-therapy are presented.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  Albumin (Low), Grade 3, n=6, 90 | 0 | 9
  Albumin (Low), Grade 4, n=6, 90 | 0 | 0
  Alkaline Phosphatase (High), Grade 3, n=6, 89 | 0 | 2
  Alkaline Phosphatase (High), Grade 4, n=6, 89 | 0 | 0
  Alanine Amino Transferase (High), Grade 3, n=6, 89 | 0 | 6
  Alanine Amino Transferase (High), Grade 4, n=6, 89 | 0 | 1
  AST (High), Grade 3, n=6, 86 | 0 | 5
  AST (High), Grade 4, n=6, 86 | 0 | 2
  Total Bilirubin (High), Grade 3, n=6, 89 | 0 | 3
  Total Bilirubin (High), Grade 4, n=6, 89 | 0 | 0
  Calcium (hypercalcemia), Grade 3, n=6, 91 | 0 | 0
  Calcium (hypercalcemia), Grade 4, n=6, 91 | 0 | 0
  Calcium (hypocalcemia), Grade 3, n=6, 91 | 0 | 8
  Calcium (hypocalcemia), Grade 4, n=6, 91 | 0 | 2
  Creatinine (High), Grade 3, n=6, 91 | 0 | 0
  Creatinine (High), Grade 4, n=6, 91 | 0 | 0
  Glucose (hyperglycemia), Grade 3, n=6, 91 | 0 | 7
  Glucose (hyperglycemia), Grade 4, n=6, 91 | 0 | 0
  Glucose (hypoglycemia), Grade 3, n=6, 91 | 0 | 0
  Glucose (hypoglycemia), Grade 4, n=6, 91 | 0 | 0
  Bicarbonate (Low), Grade 3, n=5, 82 | 0 | 0
  Bicarbonate (Low), Grade 4, n=5, 82 | 0 | 0
  Potassium (hyperkalemia), Grade 3, n=6, 91 | 0 | 1
  Potassium (hyperkalemia), Grade 4, n=6, 91 | 0 | 0
  Potassium (hypokalemia), Grade 3, n=6, 91 | 0 | 7
  Potassium (hypokalemia), Grade 4, n=6, 91 | 0 | 0
  Magnesium (hypermagnesemia), Grade 3, n=6, 88 | 0 | 3
  Magnesium (hypermagnesemia), Grade 4, n=6, 88 | 0 | 0
  Magnesium (hypomagnesemia), Grade 3, n=6, 88 | 0 | 0
  Magnesium (hypomagnesemia), Grade 4, n=6, 88 | 0 | 0
  Sodium (hypernatremia), Grade 3, n=6, 91 | 0 | 0
  Sodium (hypernatremia), Grade 4, n=6, 91 | 0 | 0
  Sodium (hyponatremia), Grade 3, n=6, 91 | 2 | 9
  Sodium (hyponatremia), Grade 4, n=6, 91 | 0 | 0
  Phosphorus, Grade 3, n=6, 88 | 0 | 5
  Phosphorus, Grade 4, n=6, 88 | 0 | 1

4. Primary Outcome: Number of Participants With a Change From Baseline in Heart Rate by Dose
Description: Change from Baseline in heart rate is categorized as decrease to <60 beats per minute (bpm), change to normal or no change, and increase to >100 bpm. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants are counted twice if the participant heart rate value decreased to <60 bpm and increased to >100 bpm post-baseline. Only those participants (par.) with heart rate values for worst-case on-therapy are presented.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  Decrease to <60, n=6, 90 | 0 | 10
  No Change, n=6, 90 | 4 | 67
  Increase to >100, n=6, 90 | 2 | 19

5. Primary Outcome: Number of Participants With a Change From Baseline in Systolic and Diastolic Blood Pressure by Dose
Description: Change from Baseline in systolic blood pressure (SBP) is categorized as: Grade 0 (<120 millimeters of mercury [mmHg]), Grade 1 (120-139 mmHg), Grade 2 (140-159 mmHg), and Grade 3/4 (>=160 mmHg). Change from Baseline in diastolic blood pressure (DBP) is categorized as: Grade 0 (<80 mmHg), Grade 1 (80-89 mmHg), Grade 2 (90-99 mmHg), and Grade 3/4 (>=100 mmHg). An increase is defined as an increase in the CTCAE grade relative to the Baseline grade. Participants with missing Baseline values are assumed to have a Baseline value of grade 0. Only those participants (par.) with blood pressure values for worst-case on-therapy are presented.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  DBP, Increase to Grade 1, n=6, 90 | 1 | 23
  DBP, Increase to Grade 2, n=6, 90 | 1 | 13
  DBP, Increase to Grade 3/4, n=6, 90 | 0 | 4
  SBP, Increase to Grade 1, n=6, 90 | 0 | 16
  SBP, Increase to Grade 2, n=6, 90 | 2 | 19
  SBP, Increase to Grade 3/4, n=6, 90 | 1 | 13

6. Primary Outcome: Number of Participants With a Change From Baseline in Temperature by Dose
Description: Change from Baseline in temperature is categorized as a decrease to <=35 degrees celsius (C), change to normal or no change, and increase to >=38 degrees C. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants (par.) are counted twice if the participant temperature value decreased to <=35 degrees C and increased to >=38 degrees C post-Baseline. Only those participants with temperature values for worst-case on-therapy are presented.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 6 | 91
Participants
  Decrease to <=35, n=6, 90 | 0 | 4
  No Change, n=6, 90 | 4 | 76
  Increase to >=38, n=6, 90 | 2 | 12

7. Primary Outcome: Number of Participants With an Investigator-assessed Best Response (Achieving Complete Response [CR], Marrow CR, Partial Response [PR], Complete Response Without Platelet Recovery [CRp] or Morphologic Leukaemia-free State[MLFS]) by Cohort
Description: Overall response rate (ORR=CR+CRp+Marrow CR+MLFS+PR) was calculated from the investigator's assessment of response recorded within the first eight weeks of treatment. CR includes complete remission. Complete remission is a state in which the participant must be free of all symptoms related to leukemia and have an absolute neutrophil count >=1 x 10^9/L, platelet count >=100 x 10^9/L, and normal marrow differential (<=5% blasts). PR includes partial remission. Partial remission is a state in which the participant has a CR with 6 to 25% abnormal cells in the marrow or 50% decrease in bone marrow blasts. CRp is as per CR but platelet count <100 x 10^9/L. MLFS is a state in which the participant has a normal marrow differential (<5% blasts), neutrophil, and platelet counts are not considered.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days)
Population: Efficacy Population: all participants included in the All Treated Population who had received at least one dose of 2 mg of study drug in Phase 2. The number of participants for the Cohort 2: AML/MDS/CMML with RAS wt/Unknown treatment group is equal to the 8 participants from Phase 1 plus the 22 participants from Phase 2 (total of 30).
Measure: Number; unit: Participants
Arm/Group | Cohort 1: AML/MDS With RAS Mutation | Cohort 2: AML/MDS/CMML With RAS wt/Unknown | Cohort 3: CMML With RAS Mutation
Number analyzed (Participants) | 50 | 30 | 11
Participants
  CR | 4 | 0 | 1
  CRp | 1 | 0 | 1
  Marrow CR | 1 | 0 | 1
  MLFS | 3 | 0 | 0
  PR | 1 | 1 | 0
  ORR | 10 | 1 | 3

8. Secondary Outcome: AUC(0-24), AUC(0-t), and AUC(0-tau) of GSK1120212 in Part 1
Description: Area under the concentration-time (AUC) curve from time zero (pre-dose) to 24 hours (AUC[0-24]) for Cycle 1 Day 1 (C1D1), from time zero to the last time of a quantifiable concentration (AUC[0-t]) for C1D1 and Cylce 1 Day 15 (C1D15) and AUC curve over the dosing interval AUC[0-tau] for C1D15 were measured. Blood samples for PK analysis were taken on Day 1 and Day 15 (within 30 minutes [min] before study drug administration) and at 0.5 hour (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 24 h post-dose. All other PK sampling were done pre-dose (i.e., within 30 min before study drug administration).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15
Population: Pharmacokinetic Population: all participants included in the All Treated Population for whom a PK sample was obtained and analyzed. Only participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter
Groups:
- GSK1120212 0.5 mg OD/ 3/1 mg LD/OD: Participants with relapsed or refractory leukemias received either GSK1120212 0.5 mg OD or 3/1 mg LD/OD as a continuous dose.
- GSK1120212 1 mg OD: Participants with relapsed or refractory leukemias received GSK1120212 1 mg OD as a continuous dose.
Arm/Group | GSK1120212 0.5 mg OD/ 3/1 mg LD/OD | GSK1120212 1 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 3 | 2 | 9
nanograms*hour/milliliter
  C1D1, AUC(0-24), n=3, 2, 9 | 77.6 (25.1) | 29.4 (5.2) | 28.0 (51.0)
  C1D1, AUC(0-t), n=3, 2, 9 | 77.6 (25.1) | 29.4 (5.2) | 28.0 (51.0)
  C1D15, AUC(0-t), n=2, 2, 8 | 172 (18.4) | 155 (61.9) | 298 (58.8)
  C1D15, AUC(0-tau), n=2, 2, 8 | 170 (17.2) | 241 (5.6) | 330 (34.6)

9. Secondary Outcome: Cmin and Cmax of GSK1120212 in Part 1
Description: Cmax is defined as the maximum observed concentration of GSK1120212 and was measured for C1D1 and C1D15. Cmin is defined as the minimal observed concentration of GSK1120212 and was measured for C1D15. Blood samples for PK analysis were taken on Day 1 and Day 15 (within 30 min before study drug administration) and at 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 24 h post-dose. All other PK sampling were done pre-dose (i.e., within 30 min before study drug administration).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15
Population: Pharmacokinetic Population. Only participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GSK1120212 0.5 mg OD/ 3/1 mg LD/OD | GSK1120212 1 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 3 | 2 | 9
nanograms per milliliter (ng/mL)
  C1D1, Cmax, n=3, 2, 9 | 7.67 (27.6) | 3.69 (35.5) | 3.27 (93.2)
  C1D15, Cmax , n=2, 2, 8 | 12.3 (19.4) | 15.1 (15.6) | 18.7 (36.1)
  C1D15, Cmin, n=2, 2, 8 | 4.79 (6.6) | 8.50 (19.4) | 10.8 (36.8)

10. Secondary Outcome: t1/2 at C1D1 and t1/2 Effective (Eff.) at C1D15 of GSK1120212 in Part 1
Description: t1/2 is defined as terminal phase half-life, which is the time required for the amount of the drug in the body to decrease by half and was measured for C1D1. t1/2eff. is defined as the effective half-life and was measured for C1D15. Blood samples for PK analysis were taken on Day 1 and Day 15 (within 30 min before study drug administration) and at 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 24 h post-dose. All other PK sampling were done pre-dose (i.e., within 30 min before study drug administration).
Time Frame: Cycle 1 Day 1 (t1/2) and Cycle 1 Day 15 (t1/2eff)
Population: Pharmacokinetic Population. Only participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK1120212 0.5 mg OD/ 3/1 mg LD/OD | GSK1120212 1 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 3 | 2 | 9
Hours
  C1D1, t1/2, n=3, 1, 8 | 33.5 (43.7) | 25.0 (NA) — There is only one participant in this cohort so dispersion can not be calculated. | 37.0 (76.2)
  C1D15, t1/2 eff., n=2, 2, 8 | 96.41 (18.1) | 128 (11.6) | 174 (80.3)

11. Secondary Outcome: Tmax of GSK1120212 in Part 1
Description: Tmax is defined as the time to reach the observed maximum concentration and was measured for C1D1 and C1D15. Blood samples for PK analysis were taken on Day 1 and Day 15 (within 30 min before study drug administration) and at 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 24 h post-dose. All other PK sampling were done pre-dose (i.e., within 30 min before study drug administration).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15
Population: Pharmacokinetic Population. Only participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK1120212 0.5 mg OD/ 3/1 mg LD/OD | GSK1120212 1 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 3 | 2 | 9
Hours
  C1D1, tmax, n=3, 2, 9 | 2.0 [1.00 to 3.00] | 1.25 [1.00 to 1.50] | 3.0 [0.50 to 5.00]
  C1D15, tmax, n=2, 2, 8 | 1.75 [1.50 to 2.00] | 2.25 [1.00 to 3.50] | 3.0 [1.00 to 24.00]

12. Secondary Outcome: Accumulation Ratio (AR) of GSK1120212 in Part 1
Description: AR is the ratio of the Day 15 AUC0-tau (0 hour to last dose interval) and Day 1 AUC0-tau (AUCtau C1D15/AUCtau C1D1). Blood samples for PK analysis were taken on Day 1 and Day 15 (within 30 min before study drug administration) and at 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, and 24 h post-dose. All other PK sampling were done pre-dose (i.e., within 30 min before study drug administration).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15
Population: Pharmacokinetic Population. Only participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | GSK1120212 0.5 mg OD/ 3/1 mg LD/OD | GSK1120212 1 mg OD | GSK1120212 2 mg OD
Number analyzed (Participants) | 2 | 2 | 8
Ratio | 6.32 (16.5) | 8.19 (10.8) | 11.1 (76.5)

13. Secondary Outcome: Ctau of GSK1120212 in Part 2
Description: Ctau is the pre-dose (trough) concentration at the end of the dosing interval and was measured for Cycle 1 Day 15 (C1D15), Cycle 2 Day 1(C2D1), Cylce 3 Day 1 (C3D1), Cycle 4 Day 1 (C4D1), Cycle 5 Day 1 (C5D1), Cycle 6 Day 1 (C6D1), Cycle 7 Day 1 (C7D1), Cycle 8 Day 1 (C8D1), Cycle 9 Day 1 (C9D1), Cycle 10 Day 1 (C10D1), Cycle 11 Day 1 (C11D1) and Cycle 12 Day 1 (C12D1). Blood samples for PK analysis were collected pre-dose (i.e., no later than 15 min prior to dosing).
Time Frame: C1D15, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1 and C12D1
Population: Pharmacokinetic Population. Only participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GSK1120212 2 mg OD
Number analyzed (Participants) | 75
nanograms per milliliter (ng/mL)
  C1D15, n=72 | 10.8 (63.8)
  C2D1, n=57 | 9.34 (78.9)
  C3D1, n=38 | 10.0 (64.9)
  C4D1, n=21 | 9.17 (99.9)
  C5D1, n=10 | 12.05 (37.4)
  C6D1, n=6 | 9.73 (44.8)
  C7D1, n=6 | 8.94 (55.0)
  C8D1, n=5 | 6.01 (222.3)
  C9D1, n=3 | 11.3 (30.7)
  C10D1, n=2 | 5.01 (73.9)
  C11D1, n=1 | 2.01 (NA) — There is only one participant in this cohort so dispersion can not be calculated.
  C12D1, n=1 | 0.644 (NA) — There is only one participant in this cohort so dispersion can not be calculated.

14. Secondary Outcome: Overall Survival by Cohort
Description: Overall survival is defined as the time from the start of study treatment (GSK1120212) until death due to any cause. For the analysis of overall survival, the last date of known contact was used for those participants who had not died at the time of analysis; such participants were considered censored.
Time Frame: From the start of the study drug until the final study visit (up to approximately 407 days )
Population: Efficacy Population. The number of participants for the Cohort 2: AML/MDS/CMML with RAS wt/Unknown treatment group is equal to the 8 participants from Phase 1 plus the 22 participants from Phase 2 (total of 30).
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: AML/MDS With RAS Mutation | Cohort 2: AML/MDS/CMML With RAS wt/Unknown | Cohort 3: CMML With RAS Mutation
Number analyzed (Participants) | 50 | 30 | 11
Months | 4.9 [4.0 to 5.7] | 3.0 [1.8 to 7.4] | 14.5 [8.6 to NA] — Due to the high censoring rate, the upper bound of the 95% CI cannot be calculated.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study drug until the final study visit (up to approximately 407 days).
Description: SAEs and non-serious AEs were collected in members of the All treated Population, comprised of all participants (par.) who received at least one dose of study medication. One Phase 2 par. was incorrectly dosed (received <2 mg [0.5 mg]); thus, 6 par. receiving GSK1120212 <2 mg OD were analyzed. .
Arm/Group | GSK1120212 <2 mg OD | GSK1120212 2 mg OD
Serious Adverse Events (participants affected / at risk) | 2/6 | 64/91
Other Adverse Events (participants affected / at risk) | 6/6 | 90/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 <2 mg OD (N=6) | GSK1120212 2 mg OD (N=91)
Pneumonia (Infections and infestations) | 1 | 17
Sepsis (Infections and infestations) | 0 | 7
Urinary tract infection (Infections and infestations) | 1 | 4
Bacteraemia (Infections and infestations) | 0 | 4
Cellulitis (Infections and infestations) | 0 | 4
Staphylococcal infection (Infections and infestations) | 0 | 3
Bacterial sepsis (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Oral infection (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Zygomycosis (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 15
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Asthenia (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 1
Graft versus host disease in intestine (Immune system disorders) | 0 | 1
Blood culture positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 <2 mg OD (N=6) | GSK1120212 2 mg OD (N=91)
Diarrhoea (Gastrointestinal disorders) | 5 | 43
Nausea (Gastrointestinal disorders) | 3 | 24
Vomiting (Gastrointestinal disorders) | 2 | 18
Constipation (Gastrointestinal disorders) | 1 | 12
Abdominal pain (Gastrointestinal disorders) | 0 | 11
Stomatitis (Gastrointestinal disorders) | 0 | 7
Gingival bleeding (Gastrointestinal disorders) | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 5
Oral pain (Gastrointestinal disorders) | 1 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 22
Oedema peripheral (General disorders) | 3 | 21
Pyrexia (General disorders) | 3 | 21
Mucosal inflammation (General disorders) | 0 | 9
Asthenia (General disorders) | 0 | 6
Chills (General disorders) | 0 | 5
Pain (General disorders) | 1 | 2
Swelling (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 6
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 13
Decreased appetite (Metabolism and nutrition disorders) | 2 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 11
Urinary tract infection (Infections and infestations) | 2 | 10
Cellulitis (Infections and infestations) | 0 | 8
Staphylococcal infection (Infections and infestations) | 1 | 6
Enterococcal infection (Infections and infestations) | 1 | 2
Gingivitis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 1
Vulval cellulitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 21
Aspartate aminotransferase increased (Investigations) | 2 | 19
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Brain natriuretic peptide increased (Investigations) | 1 | 1
Prothrombin time prolonged (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 10
Dizziness (Nervous system disorders) | 1 | 4
Syncope (Nervous system disorders) | 0 | 5
Presyncope (Nervous system disorders) | 1 | 1
Vision blurred (Eye disorders) | 2 | 13
Glaucoma (Eye disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 7
Tachycardia (Cardiac disorders) | 1 | 7
Pericardial effusion (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 5
Haematuria (Renal and urinary disorders) | 0 | 5
Renal failure acute (Renal and urinary disorders) | 1 | 4
Dysuria (Renal and urinary disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 7
Haematoma (Vascular disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 6
Insomnia (Psychiatric disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.